CLINICAL TRIAL: NCT01522859
Title: The Efficacy of Telehealth Monitoring in the Management of Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Telehealth Monitoring in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Eastern Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, JE McDowell, Principal Investigator, South Eastern Health and Social Care Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09/NIR01/26
Record Dates: First submitted 2012-01-24; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Telehealth; health related quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard care (No Intervention): A standardised home based programme of specialist respiratory assessment and monitoring provided by the local Community Respiratory Team (CRT) and General Practitioner (GP) for a period of six months.
- Telehealth monitoring (Experimental): Daily monitoring of patient's health status using a small telecommunications device.
  Interventions: Device: Telehealth monitoring system (Honni Med)

INTERVENTIONS:
Device: Telehealth monitoring system (Honni Med) — The system is uploaded with personal information including: monitoring start time; clinical observations (blood pressure, heart rate, oxygen saturations); and questions relating to symptoms. The patient is instructed on use and observed monitoring. The patient is monitored daily for a period of six months. The monitoring session lasts approximately 10 minutes during which the patient attaches a finger probe and blood pressure cuff and responds 'yes' or 'no' to the set questions. Daily data is transmitted via a phone line to a secure server to be downloaded and reviewed by a Telehealth nurse.If one or more of the clinical observations is outside normal limits the appropriate healthcare intervention is utilised.
  Other Names: Honni Med
  Arms: Telehealth monitoring

SUMMARY:
The the aim of this study is to determine the benefits of Telehealth monitoring in the management of patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major burden on healthcare systems worldwide. The current management of patients with COPD includes well established interventions such as pulmonary rehabilitation and inhaled therapies which have demonstrated variable impact on reducing rates of exacerbation and improving health related quality of life.

Telehealth is a home monitoring system used to record clinical observations and carry out question and answer sessions. It has been proposed that Telehealth medicine may offer an alternative strategy to the overall management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of moderate to severe chronic obstructive pulmonary disease (COPD)
* a minimum of two: Emergency Department admissions; hospital admissions or emergency GP contacts in the 12 months previous to the study

Exclusion Criteria:

* any respiratory disorder other than COPD
* patients cognitively unable to learn the process of monitoring

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in St Georges's Respiratory Questionnaire at six months | Baseline and six months
  Self completed questionnaire

SECONDARY OUTCOMES:
Change from baseline in EuroQol at six months | Baseline and six months
  self completed questionnaire
Change from baseline in Hospital Anxiety and Depression Scale at six months | Baseline and six months
  self administered questionnaire
healthcare utilisation | six months
  data collected retrospectively from healthcare notes and hospital coding
number of exacerbations | six months
  data collected retrospectively from healthcare notes
satisfaction | six months
  interview administered questionnaire
cost effectiveness | six months
  QALY analysis

CONTACTS AND LOCATIONS:
Overall Officials: Janet E McDowell, BScHons, PhD, Principal Investigator — South Eastern Health and Social Care Trust; Stephen Tate, BSc,MD,FRCP, Study Director — South Eastern Health and Social Care Trust
Locations (1):
- South Eastern Health and Social Care Trust, Lisburn, Co Antrim, United Kingdom